CLINICAL TRIAL: NCT04184284
Title: imPROve-asthma - A Prospective, 24-month, Observational Study to Investigate the Change in Patient-Reported Outcomes in Severe Eosinophilic Asthma Patients Treated With Benralizumab Biologic Therapy Under Real-life Conditions in Germany
Brief Title: Change in Patient-Reported Outcomes in Severe Eosinophilic Asthma Patients Treated With Benralizumab Under Real-life Conditions
Acronym: imPROve
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3250R00053
Record Dates: First submitted 2019-10-13; First posted 2019-12-03 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Asthma
Keywords: benralizumab
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Primary Study Cohort - Anti-IL5/IL5R naïve patients: Severe eosinophilic asthma patients who have never received anti-Interleukin-5 / anti-Interleukin-5-receptor (anti-IL-5/anti-IL-5R) biologic treatment for severe eosinophilic asthma, for whom the investigator had decided to initiate benralizumab biologic treatment.
- Secondary Study Cohort - Biologic experienced patients: Patients that previously received a biologic treatment for severe asthma (at least one dose).

SUMMARY:
The main aim of this study is to investigate the change in asthma control after 6 months of therapy in patients treated with benralizumab biologic therapy for severe eosinophilic asthma under real-life conditions in a pulmonary care setting in Germany. The study also aims to investigate Quality-of-Life (QoL), the early treatment response, treatment effectiveness and the change in asthma control over time, following benralizumab therapy. This study will also describe the physician-chosen reasons for starting beralizumab therapy or switching to benralizumab therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 years or older with confirmed diagnosis of severe asthma according to the ATS/ERS and local German guidelines
* Decision was made by the investigator (regardless of this NIS) to start treating the patient with benralizumab according to severe eosinophilic asthma indication (NB: can include patients that are switched from another EU approved biologic treatment if required for a medical reason).
* Patients must be able and willing to read and comprehend written instructions, and comprehend and complete the questionnaires required by the protocol
* After full explanation, patients must have signed an informed consent document indicating that they understand the purpose of and the procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

* Concomitant treatment with any other biologic for any indication
* Patients already treated with benralizumab
* Clinically important pulmonary disease other than asthma including: chronic obstructive pulmonary disease (as main diagnosis), bronchiectasis, idiopathic pulmonary fibrosis, pulmonary hypertension, alpha-1-antitrypsin-deficiency, and malignancy of any kind (NB: the following conditions are permitted: nasal polyposis, allergic rhinitis, atopic dermatitis, non-idiopathic pulmonary fibrosis).
* An acute or chronic condition that, in the investigator's opinion, would limit the patient's ability to complete questionnaires or participate in this study or impact the interpretations of results.
* Concurrent biologics for asthma are not allowed except for stable allergen immunotherapy (defined as a stable dose and regimen at the time of enrolment). Acceptable wash-out periods for other asthma biologics: ≥30 days from last dose of previous biologic
* Pregnancy or lactation period
* Participation in an observational trial that might, in the investigator's opinion, influence the assessment for the current study, or participation in a randomized clinical trial in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: approximately 350 to 500 patients in 70 pulmonology sites (hospitals and outpatient practices) in Germany Primary study cohort: approximately 250 patients Secondary study cohort: approximately 100 to 250 patients
Sampling Method: Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
The change in asthma control after 6 months of treatment in anti-IL5/IL5R naïve patients initiated with benralizumab treatment | Baseline and 6 months after baseline
  Change from baseline in (Asthma Control Test - questionnaire) ACT score after 6 months treatment in anti-IL5/IL5R naïve patients. ACT is a simple, validated, 5-item tool giving a total score from 5 (worst control) to 25 (best control). Scores of 20 to 25 denote well-controlled asthma, scores ≤19 identifies patients with poorly controlled asthma. The minimum clinically important difference (MCID) is reported to be 3 points.

SECONDARY OUTCOMES:
The investigator reported treatment effectiveness after 6 months of treatment in anti-IL5/IL5R naïve patients initiated with benralizumab treatment | 6 months after first treatment
  Investigator-reported treatment effectiveness using GETE (Global Evaluation of Treatment Effectiveness) after 6 months of treatment. GETE grades overall treatment effectiveness using the following criteria: excellent (complete control of asthma); good (marked improvement of asthma); moderate (discernible, but limited improvement in asthma); poor (no appreciable change in asthma); or worsening (of asthma).
The change in health-related quality of life (HRQL) in anti-IL5/IL5R naïve patients initiated with benralizumab treatment | Baseline and 6 months after first treatment
  Change from baseline in St. George's Respiratory Questionnaire (SGRQ) total score and domain scores (symptoms, activity and impact score) after 6 months treatment in anti-IL5/IL5R naïve patients. SGRQ is a validated, 50-item questionnaire, giving scores ranging from 0 (best health status) to 100 (worst health status). The SGRQ yields a total score and 3 domain scores (symptoms, activity, and impacts). The total score indicates the impact of disease on overall health status. A difference of four units in the SGRQ total score is considered the MCID.
The early treatment response in anti-IL5/IL5R naïve patients initiated with benralizumab treatment, day 7, ACQ-6 | Baseline and day 7 after first treatment
  Change from baseline in ACQ-6 (Asthma-Control-Questionnaire-6) score after 7 days of treatment in anti-IL5/IL5R naïve patients.
  ACQ-6 is a validated questionnaire based on 5 symptoms questions (night-time waking, symptoms on waking, activity limitation, shortness of breath, wheezing), and daily rescue bronchodilator use. Each item is scored on a 7-point scale (0=no impairment; 6=maximum impairment), and the ACQ score is the mean of these items. The MCID is greater than or equal to 0.5.
The early treatment response in anti-IL5/IL5R naïve patients initiated with benralizumab treatment, day 7, VAS-1 | Baseline and day 7 after first treatment
  Change from baseline in patient satisfaction, measured on Visual Analogue Scale (VAS), after 7 days of treatment in anti-IL5/IL5R naïve patients. VAS Scores ranged from "extremly satisfied" (0 mm) to "not at all satisfied" (100 mm).
The early treatment response in anti-IL5/IL5R naïve patients initiated with benralizumab treatment, day 7, VAS-2 | Baseline and day 7 after first treatment
  Change from baseline in patient symptoms, measured on Visual Analogue Scale (VAS), after 7 days of treatment in anti-IL5/IL5R naïve patients. VAS Scores ranged from "not at all bothersome" (0 mm) to "extremly bothersome" (100 mm).
The early treatment response in anti-IL5/IL5R naïve patients initiated with benralizumab treatment, day 14, ACQ-6 | Baseline and day 14 after first treatment
  Change from baseline in ACQ-6 (Asthma-Control-Questionnaire-6) score after 14 days of treatment in anti-IL5/IL5R naïve patients. ACQ-6 is a validated questionnaire based on 5 symptoms questions (night-time waking, symptoms on waking, activity limitation, shortness of breath, wheezing), and daily rescue bronchodilator use. Each item is scored on a 7-point scale (0=no impairment; 6=maximum impairment), and the ACQ score is the mean of these items. The MCID is greater than or equal to 0.5.
The early treatment response in anti-IL5/IL5R naïve patients initiated with benralizumab treatment, day 14, VAS-1 | Baseline and day 14 after first treatment
  Change from baseline in patient satisfaction, measured on Visual Analogue Scale (VAS), after 14 days of treatment in anti-IL5/IL5R naïve patients. VAS Scores ranged from "extremly satisfied" (0 mm) to "not at all satisfied" (100 mm).
The early treatment response in anti-IL5/IL5R naïve patients initiated with benralizumab treatment, day 14, VAS-2 | Baseline and day 14 after first treatment
  Change from baseline in patient symptoms, measured on Visual Analogue Scale (VAS), after 14 days of treatment in anti-IL5/IL5R naïve patients. VAS Scores ranged from "not at all bothersome" (0 mm) to "extremly bothersome" (100 mm).
The change of asthma control over time and the maintained response after initiation of benralizumab treatment in anti-IL5/IL5R naïve patients initiated with benralizumab treatment using ACT | Date of enrollment until end of follow-up (approx. 24 months after enrollment)
  Change from baseline in asthma control at each visit during the study period, using ACT in anti-IL5/IL5R naïve patients. ACT is a simple, validated, 5- item tool giving a total score from 5 (worst control) to 25 (best control). Scores of 20 to 25 denote well-controlled asthma, scores ≤19 identifies patients with poorly controlled asthma. The minimum clinically important difference (MCID) is reported to be 3 points.
The change of asthma control over time and the maintained response after initiation of benralizumab treatment in anti-IL5/IL5R naïve patients initiated with benralizumab treatment using ACQ-6 | Date of enrollment until end of follow-up (approx. 24 months after enrollment)
  Change from baseline in asthma control at each visit during the study period, using ACQ-6 in anti-IL5/IL5R naïve patients. ACQ-6 is a validated questionnaire based on 5 symptoms questions (night-time waking, symptoms on waking, activity limitation, shortness of breath, wheezing), and daily rescue bronchodilator use. Each item is scored on a 7-point scale (0=no impairment; 6=maximum impairment), and the ACQ score is the mean of these items. The MCID is greater than or equal to 0.5.
The reasons for biologic treatment change | Date of enrollment until end of follow-up (approx. 24 months after enrollment)
  Investigator-chosen reasons for
  * Initiation of benralizumab / switching to benralizumab (treatment change from one biologic to another, regardless of the time since the last dose of the previous biologic) at enrolment
  * discontinuation of benralizumab during the treatment period.

OTHER OUTCOMES:
The change of physical activity over time in anti-IL5/IL5R naïve patients | Baseline until end of follow-up (approx. 24 months after enrollment)
  Change from baseline in steps per day over 24 months of treatment in anti-IL5/IL5R naïve patients.
The change in asthma control after 6, 12, 18 and 24 months of treatment in biologic experienced patients, using ACT | Baseline, 6, 12, 18 and 24 months after first treatment
  Change from baseline in (Asthma Control Test - questionnaire) ACT score at the end of 6, 12, 18 and 24 months of benralizumab treatment in biologic experienced patients. ACT is a simple, validated, 5-item tool giving a total score from 5 (worst control) to 25 (best control). Scores of 20 to 25 denote well-controlled asthma, scores ≤19 identifies patients with poorly controlled asthma. The minimum clinically important difference (MCID) is reported to be 3 points.
The change in asthma control and the maintained response after initiation of benralizumab treatment in biologic experienced patients using ACQ-6 | Baseline, 6, 12, 18 and 24 months after first treatment
  Change from baseline in ACQ-6 (Asthma-Control-Questionnaire-6) score at the end of 6, 12, 18 and 24 months of benralizumab treatment in biologic experienced patients.
  ACQ-6 is a validated questionnaire based on 5 symptoms questions (night-time waking, symptoms on waking, activity limitation, shortness of breath, wheezing), and daily rescue bronchodilator use. Each item is scored on a 7-point scale (0=no impairment; 6=maximum impairment), and the ACQ score is the mean of these items. The MCID is greater than or equal to 0.5.
The change in HRQL after 6, 12, 18 and 24 months of treatment in biologic experienced patients | Baseline, 6, 12, 18 and 24 months after first treatment
  Change from baseline in St. George's Respiratory Questionnaire (SGRQ) total score and domain scores (symptoms, activity and impact score) after 6, 12, 18 and 24 months treatment in biologic experienced patients. SGRQ is a validated, 50-item questionnaire, giving scores ranging from 0 (best health status) to 100 (worst health status). The SGRQ yields a total score and 3 domain scores (symptoms, activity, and impacts). The total score indicates the impact of disease on overall health status. A difference of four units in the SGRQ total score is considered the MCID.
The early treatment response in biologic experienced patients initiated with benralizumab treatment, ACQ-6 | Baseline, day 7 and day 14 after first treatment
  Change from baseline in ACQ-6 (Asthma-Control-Questionnaire-6) score after 7 and 14 days of treatment in biologic experienced patients. ACQ-6 is a validated questionnaire based on 5 symptoms questions (night-time waking, symptoms on waking, activity limitation, shortness of breath, wheezing), and daily rescue bronchodilator use. Each item is scored on a 7-point scale (0=no impairment; 6=maximum impairment), and the ACQ score is the mean of these items. The MCID is greater than or equal to 0.5.
The early treatment response in biologic experienced patients initiated with benralizumab treatment, patient satisfaction, VAS-1 | Baseline, day 7 and day 14 after first treatment
  Change from baseline in patient satisfaction, measured on Visual Analogue Scale (VAS), after 7 and 14 days of treatment in biologic experienced patients. VAS Scores ranged from "extremly satisfied" (0 mm) to "not at all satisfied" (100 mm).
The early treatment response in biologic experienced patients initiated with benralizumab treatment, patient symptoms, VAS-2 | Baseline, day 7 and day 14 after first treatment
  Change from baseline in patient symptoms, measured on Visual Analogue Scale (VAS), after 7 and 14 days of treatment in biologic experienced patients. VAS Scores ranged from "not at all bothersome" (0 mm) to "extremly bothersome" (100 mm).
The investigator reported treatment effectiveness after 6 months of treatment in biologic experienced patients initiated with benralizumab treatment | 6 months after first treatment
  Investigator-reported treatment effectiveness using GETE (Global Evaluation of Treatment Effectiveness) after 6 months of treatment. GETE grades overall treatment effectiveness using the following criteria: excellent (complete control of asthma); good (marked improvement of asthma); moderate (discernible, but limited improvement in asthma); poor (no appreciable change in asthma); or worsening (of asthma).

CONTACTS AND LOCATIONS:
Locations (50):
- Germany (50):
  - Research Site, Aschaffenburg
  - Research Site, Augsburg
  - Research Site, Bamberg
  - Research Site, Beelitz
  - Research Site, Berlin
  - Research Site, Biberach
  - Research Site, Bonn
  - Research Site, Bremen
  - Research Site, Cottbus
  - Research Site, Darmstadt
  - Research Site, Dresden
  - Research Site, Düsseldorf
  - Research Site, Flensburg
  - Research Site, Frankfurt
  - Research Site, Fürstenwalde
  - Research Site, Gelsenkirchen
  - Research Site, Gerlingen
  - Research Site, Gotingen
  - Research Site, Halberstadt
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Hemer
  - Research Site, Hettstedt
  - Research Site, Ibbenbueren
  - Research Site, Immenhausen
  - Research Site, Konstanz
  - Research Site, Leipzig
  - Research Site, Magdeburg
  - Research Site, Marburg
  - Research Site, Markkleeberg
  - Research Site, München
  - Research Site, Neu-Isenburg
  - Research Site, Peine
  - Research Site, Radebeul
  - Research Site, Regensburg
  - Research Site, Reinfeld
  - Research Site, Rheine
  - Research Site, Rostock
  - Research Site, Roth
  - Research Site, Saalfeld
  - Research Site, Schleswig
  - Research Site, Teuchern
  - Research Site, Treuenbrietzen
  - Research Site, Waren
  - Research Site, Warendorf
  - Research Site, Wedel
  - Research Site, Wiesbaden
  - Research Site, Witten

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250R00053&attachmentIdentifier=9e610f4f-74eb-4fa3-9d76-16af3879d0a4&fileName=D3250R00053_imPROve_CSR-Synopsis_V1.0_ctt_redacted.pdf&versionIdentifier=